CLINICAL TRIAL: NCT00920049
Title: Preventing Motor Vehicle Crashes Among Young Drivers: Evaluation of the AAA Checkpoints Program
Brief Title: Preventing Motor Vehicle Crashes Among Young Drivers: Evaluation of the Checkpoints Program Presented by the American Automobile Association
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 999909165; 09-CH-N165
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-29

CONDITIONS: Injury
Keywords: Driving; Injury; Prevention; Intervention; Parents
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Behavioral: Persuasion

SUMMARY:
Background:

* Automobile crash risks are highest right after licensure and decline rapidly for about 6 months and then gradually for years, regardless of the amount of supervised practice driving or age at licensure. The only approaches to this problem that have demonstrated effectiveness are Graduated Driver Licensing (GDL) and parental management.
* The Checkpoints Program consists of persuasive messages and materials designed to increase adoption of the Checkpoints Parent-Teen Driving Agreement and to improve parents' ability to set limits on higher-risk driving privileges for novice drivers. Researchers are interested in determining whether expanding the Checkpoints Program to an online version (instead of through the mail) can help improve parent limit-setting in connection with the program.

Objectives:

* To determine the feasibility and effectiveness of conducting an online version of the Checkpoints Program through American Automobile Association (AAA) clubs.
* To test rates of parental intervention and limit-setting after participation in the Checkpoints Program.

Eligibility:

- Parents whose teenage children are enrolled in AAA-affiliated driving schools.

Design:

* Parents with children at the permit stage of driver's education will be recruited through AAA clubs and will be asked to visit a designated Web site to sign up for the program.
* Parents will provide consent and complete the baseline survey, and will be assigned to random groups to test different versions of the Checkpoints Program (the intervention or a control group Web site).
* The intervention program will contain videos, regular e-mails, and newsletters on setting parental limits and information on specific teen driving risks. The control program will provide information on various topics related to the licensing procedure and safe driving, but no specific information on teen driving risks.
* A follow-up assessment will be conducted 1 month after the teenager receives his or her license.

DETAILED DESCRIPTION:
Crash risks are highest right after licensure and decline rapidly for about 6 months and then gradually for years, regardless of the amount of supervised practice driving or age at licensure. Graduate Driver Licensing (GDL) and parental management are the only approaches to this problem with demonstrated effectiveness. The Checkpoints Program consists of persuasive messages and materials designed to increase adoption of the Checkpoints Parent-Teen Driving Agreement and increase parent limit setting on higher-risk driving privileges among novice teenage drivers. The current study builds on the results of several previous trials of the Checkpoints Program that have shown significant treatment group effects on parent limit setting, teen risky driving, and violations. The purpose of this study is to determine the efficacy of conducting an online adaptation of the Checkpoints Program through the American Automobile Association (AAA) clubs. The study will be conducted with parents whose teenage children are enrolled in AAA-affiliated driving schools. 800 families will be recruited through AAA Clubs, assigned to intervention or comparison groups, provided online access to Checkpoints or comparison materials, and assessed at baseline and after teen licensure.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. The adolescent is between the ages of 15 years 6 months to 17 years 0 month at time of recruitment;
  2. The adolescent lives with the parent or legal guardian at least 50% of the time;
  3. The parent has routine access to the internet and is able to complete on line surveys in English;
  4. A parent or legal guardian agrees to participate.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2009-06-05; Primary Completion 2012-03-29 (Actual); Study Completion 2012-03-29 (Actual)

PRIMARY OUTCOMES:
Improvements in risky driving and crash risk

SECONDARY OUTCOMES:
Adoption of parent-teen driving agreement and adherence to graduated driver licensing policy

CONTACTS AND LOCATIONS:
Overall Officials: Germaine M Louis, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arnett JJ. Developmental sources of crash risk in young drivers. Inj Prev. 2002 Sep;8 Suppl 2(Suppl 2):ii17-21; discussion ii21-3. doi: 10.1136/ip.8.suppl_2.ii17. PMID 12221026
- [Background] Foss R, Goodwin A. Enhancing the effectiveness of graduated driver licensing legislation. J Safety Res. 2003 Jan;34(1):79-84. doi: 10.1016/s0022-4375(02)00083-x. PMID 12535909
- [Background] Hartos JL, Nissen WJ, Simons-Morton BG. Acceptability of the Checkpoints Parent-Teen Driving Agreement: pilot test. Am J Prev Med. 2001 Aug;21(2):138-41. doi: 10.1016/s0749-3797(01)00330-0. PMID 11457634